CLINICAL TRIAL: NCT03714438
Title: Effect of Acute Administration of Medicago Sativa on Glucose Tolerance, Insulin Secretion and Insulin Sensitivity in Normoglycemic, Overweight Adults
Brief Title: Effect of Medicago Sativa on Oral Glucose Tolerance in Healthy Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Lizet Yadira Rosales Rivera, Researcher Professor, University of Guadalajara
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CT-MS-LYZ
Record Dates: First submitted 2018-05-10; First posted 2018-10-22 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Glucose Tolerance
Keywords: Medicago sativa; Insulin secretion; Insulin Sensitivity
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medicago sativa (Experimental): 1,500 mg unique dose, 30 min before the oral glucose tolerance test.
  Interventions: Drug: Medicago Sativa
- Placebo (Placebo Comparator): 1,500 mg unique dose, 30 min before the oral glucose tolerance test.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Drug: Medicago Sativa — Single oral doses of Medicago sativa (1,500 mg), 30 min before before the oral glucose tolerance test.
  Other Names: Alfalfa; Lucerne
  Arms: Medicago sativa
Dietary Supplement: Placebo — Single oral doses of placebo (1,500 mg), 30 min before before the oral glucose tolerance test.
  Arms: Placebo

SUMMARY:
Previous preclinical investigations have found that Medicago sativa promotes the decrease of glucose concentrations. To evaluate the acute effect of Medicago sativa administration on glucose tolerance, insulin secretion, and insulin sensitivity in healthy individuals.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled, two-period, cross-over clinical trail will be carrie out in 15 healthy, sedentary individuals of both genders, who meet the following inclusion criteria: 25 to 40 years of age, normal fasting plasma glucose (≤ 5.5 mm/L), blood pressure (<130/90 mmHg), body mass index of 25 to 29.9 kg/m2, no taking any medication known to affect glucose tolerance, nondrinkers and nonsmokers. No pregnant, and lactation estate for female participants. They will be select from the same neighborhood and socioeconomic status.

After a fasting blood sample patients will be assigned at random-order through a closed-envelope selection, to receive one of two possible sequences during which they received either single oral doses of Medicago sativa or homologated placebo in 1,500 mg and were crossover with a difference of at least 7 days washout interval. Thirty minutes after each intervention patients underwent a 75-g oral glucose tolerant test (OGTT). Area under the curve of glucose and insulin, phases of insulin secretion, and insulin sensitivity will be calculate for each treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Fasting plasma glucose ≤99 mg/dL.
* Two hours postload plasma glucose (100 a 139 mg/dL).
* Body mass Index: 25 -39.9 kg/m2.
* body weight stable over the last 3 months.
* Women in follicular phase of the menstrual cycle (days 3 to 8 of the cycle) at the time of laboratory tests.
* Sedentary.
* Nonsmokers.
* Body weight unchanged upper to 5% for at least 3 moths before the study.

Exclusion Criteria:

* Women in pregnancy and/or breastfeeding
* Physical or mental disability that makes it impossible to perform the intervention.
* Diagnosis of hypertension or heart failure.
* Untreated thyroid disease.
* Consumption of oral agents or other medications or supplements with proven properties that modify the behavior of glucose and lipids (oral hypoglycemic agents, insulin, lipid-lowering).
* Diagnosis of liver disease or elevation twice of the upper normal value of liver enzymes.
* Diagnosis of renal disease or creatinine >1.5 mg/dL.
* Diagnosis of prediabetes: Fasting plasma glucose ≥100 mg/dL and/or 2h-OGTT ≥140mg/dL and/or glycated hemoglobin A1c (A1C) between 5.7 - 6-4 %.
* Diagnosis of Type 2 Diabetes Mellitus (T2DM): Fasting glucose ≥ 126 mg / dL and/or 2h-OGTT ≥ 200 mg/dL .
* Total Cholesterol ≥ 280 mg/dL.
* Triglycerides ≥ 300 mg/dL.
* Known allergy to calcined magnesia or Medicago sativa.

Ages: 30 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2017-02-07 (Actual); Primary Completion 2018-01-11 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Fasting plasma glucose (FPG) | After the acute administration of placebo and Medicago sativa. 15 days wash period between them.
  Glucose concentration after overnight fasting (10 to 12-h) determined by spectrophotometry methods. Expressed in mmol/L.
2 hour oral glucose tolerance test (2h-PG) | After the acute administration of placebo and Medicago sativa. 15 days wash period between them.
  Glucose concentration after 75-g oral dextrose load, determined by spectrophotometry methods. Expressed in mmol/L
First Phase of Insulin Secretion | After the acute administration of placebo and Medicago sativa. 15 days wash period between them.
  calculated as 1283 + 1.829 x insulin 30' (mmol/L) - 138.7 x glucose 30' + 3.772 x insulin 0' (pmol/L).
Total Insulin Secretion | After the acute administration of placebo and Medicago sativa. 15 days wash period between them.
  Insulinogenic index calculated as ΔAUC insulin /(ΔAUC glucose
Insulin sensitivity | After the acute administration of placebo and Medicago sativa. 15 days wash period between them.
  Matsuda index (insulin sensitivity) calculated as [10,000/square root of (glucose 0' X insulin 0')] (mean glucose X mean insulin during 2h-OGTT)]

SECONDARY OUTCOMES:
Body Weight | At baseline of the study
  Measured with minimal clothing and bare feet
Body Mass Index (BMI) | At baseline of the study
  Calculated with the Quetelet index
Waist circumference (WC) | At baseline of the study
  Measured with a flexible tape in them id point between the lowest rib and the iliac crest and is expressed in centimeters.
Systolic blood pressure (SBP) | At baseline of the study
  Evaluated with a digital sphygmomanometer with the subject sited down on a chair after a resting period of 5 minutes on three occasions. The mean of the three measures was considered as the value of systolic blood pressure expressed on mmHg
Diastolic Blood pressure (DBP) | At baseline of the study
  Evaluated with a digital sphygmomanometer with the subject sited down on a chair after a resting period of 5 minutes on three occasions. The mean of the three measures was considered as the value of diastolic blood pressure expressed on mmHg
Total Cholesterol (TC) | At baseline of the study
  Determined after overnight fasting (10 to 12-h), determined by spectrophotometric methods. Expressed in mmol/L.
Triglycerides (TG) | At baseline of the study
  Determined after overnight fasting (10 to 12-h), evaluated by colorimetric method, expressed on mmol/L.
High Density Lipoprotein Cholesterol (HDL- C) | At baseline of the study
  Determined after overnight fasting (10 to 12-h), evaluated by colorimetric method, expressed on mmol/L.
Low Density Lipoprotein Cholesterol (LDL-C) | At baseline of the study
  Determined after overnight fasting (10 to 12-h), calculated with the Friedewald equation LDL-C (mmol/L) = TC (mmol/L) - HDL-C (mmol/L) - [TG (mmol/L)/2.2] and very low-density lipoprotein (VLDL) for the proportion of TG (mmol/L)/2.2. Expressed in mmol/L.
Very Low Density Lipoprotein (VLDL) | At baseline of the study
  Estimated by standardized techniques
Levels of aspartate aminotransferase in blood | At baseline of the study
  Estimated by standardized techniques
Levels of alanine aminotransferase in blood | At baseline of the study
  Estimated by standardized techniques
Levels of creatinine in blood | At baseline of the study
  Estimated by standardized techniques
Levels of uric acid in blood | At baseline of the study
  Estimated by standardized techniques

CONTACTS AND LOCATIONS:
Overall Officials: Lizet Yadira Rosales-Rivera, PhD Science, Principal Investigator — Institute of Experimental and Clinical Therapeutics (INTEC), CUCS, University of Guadalajara
Locations (1):
- Institute of Experimental and Clinical Therapeutics (INTEC), CUCS, University of Guadalajara, Guadalajara, Jalisco, Mexico

REFERENCES:
- [Background] Abdul-Ghani M, DeFronzo RA, Jayyousi A. Prediabetes and risk of diabetes and associated complications: impaired fasting glucose versus impaired glucose tolerance: does it matter? Curr Opin Clin Nutr Metab Care. 2016 Sep;19(5):394-399. doi: 10.1097/MCO.0000000000000307. PMID 27389083
- [Background] Gawel E. Chemical composition of lucerne leaf extract (EFL) and its applications as a phytobiotic in human nutrition. Acta Sci Pol Technol Aliment. 2012 Jul-Sep;11(3):303-10. PMID 22744951
- [Background] Tai MM. A mathematical model for the determination of total area under glucose tolerance and other metabolic curves. Diabetes Care. 1994 Feb;17(2):152-4. doi: 10.2337/diacare.17.2.152. PMID 8137688
- [Background] Stumvoll M, Mitrakou A, Pimenta W, Jenssen T, Yki-Jarvinen H, Van Haeften T, Renn W, Gerich J. Use of the oral glucose tolerance test to assess insulin release and insulin sensitivity. Diabetes Care. 2000 Mar;23(3):295-301. doi: 10.2337/diacare.23.3.295. PMID 10868854